CLINICAL TRIAL: NCT06437210
Title: Evaluation of Treatment With Viusid in Post-COVID-19 Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIUSID_POSTCOVID_CO_2022
Record Dates: First submitted 2024-05-30; First posted 2024-05-31 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Post-COVID-19 Syndrome; COVID-19; Dyspnea; Fatigue; Cough; Inflammation
Keywords: COVID-19; Antioxidants; Post-COVID-19 Syndrome; Fatigue; Immunomodulator
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19; Dyspnea; Fatigue; Cough; Inflammation | interventions — Viusid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Viusid Group (Experimental): Oral administration of viusid oral solution 30 mL 3 times a day with the main meals (breakfast, lunch and dinner) for 30 days.
  Interventions: Dietary Supplement: Viusid Oral Solution
- Placebo Group (Placebo Comparator): Oral administration of placebo 30 mL 3 times a day with the main meals (breakfast, lunch and dinner) for 30 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Viusid Oral Solution — Patients in the experimental intervention group will be administered Viusid Oral Solution (CATALYSIS S.L., Madrid, Spain) 30 mL orally 3 times a day with the main meals (breakfast, lunch and dinner) for 30 days.
  Arms: Viusid Group
Dietary Supplement: Placebo — Patients in the experimental intervention group will be administered Placebo (CATALYSIS S.L., Madrid, Spain) 30 mL orally 3 times a day with the main meals (breakfast, lunch and dinner) for 30 days.
  Arms: Placebo Group

SUMMARY:
Reports of long-lasting symptoms of COVID-19 are increasing, but little is known about the prevalence of risk factors or whether it is possible to predict a prolonged course at disease onset. Prolonged COVID is characterized on the basis of symptoms such as fatigue, headache, dyspnea, and anosmia present for weeks, with older age, high body mass index, and female sex being more susceptible.

Accordingly, and in the absence of specific treatments, the present study seeks to establish a treatment protocol for Post-COVID syndrome through the application of the dietary supplement VIUSID, due to its anti-inflammatory and immunomodulatory effect, thus helping to reduce and/or control the symptoms of the syndrome.

DETAILED DESCRIPTION:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2e) is the pathogen responsible for the 2019 coronavirus disease pandemic (COVID-19), which has caused global health care crises and overstretched health care resources, Scientific and clinical evidence is evolving on the subacute and long-term effects of COVID-19, which can affect multiple organ systems. As the population of patients recovering from COVID-19 grows, it is critical to establish an understanding of the healthcare issues surrounding them. COVID-19 is now recognized as a multi-organ disease with a broad spectrum of manifestations.

Early reports suggest residual effects of SARS-CoV-2c infection, such as fatigue, dyspnea, chest pain, cognitive impairment, arthralgia and impaired quality of life. Cellular damage, a robust innate immune response with inflammatory cytokine production and a procoagulant state induced by SARS-CoV-2 infection may contribute to these sequelae. Survivors of previous coronavirus infections, including the 2003 SARS epidemic and the 2012 Middle East Respiratory Syndrome (MERS) outbreak, have demonstrated a similar set of persistent symptoms, reinforcing concerns about clinically significant sequelae of COVID-19.

Some countries use several drugs to treat coronavirus. In one of its documents, the Spanish Society of Medicine mentions the recommendations of the protocol developed for the treatment of COVID-19. Specific antiviral treatment requires drugs such as lopinavir/ritonavir administered orally. This drug is indicated to help control human immunodeficiency virus (HIV) infection. It is only administered orally 0 in concomitant treatment with interferon beta-lb. In this case Betaferon is recommended, which is indicated for the treatment of multiple sclerosis. Interferons are proteins produced by the body that help fight against attacks on the immune system, such as viral infections. Lopinavir / ritonavir can also be used in combination with an alpha-2B interferon, such as Intron A, which modifies the immune system response of the patient. the body's immune system to help fight infections and serious illnesses.

Viusid (Catalysis Laboratories, Madrid, Spain) is a nutritional supplement with recognized antioxidant and immunomodulatory properties that have beneficial effects on clinical outcomes related to cirrhosis, such as survival, disease progression and the development of hepatocellular carcinoma (HCC). It contains different molecules (ascorbic acid, zinc and glycyrrhizic acid) with recognized antioxidant and immunomodulatory properties. Glycyrrhizin (0.033g), the most important active ingredient of the supplement, is known to have an immunomodulatory, antiviral and biological effect, and has also demonstrated various anti-inflammatory properties (such as increased production of IL-10: a potent anti-inflammatory cytokine that inhibits the synthesis of many proinflammatory proteins), as well as an anti-apoptotic effect, hepatocyte proliferation and stabilization of cell membranes in the liver. Recent data suggest that Viusid ameliorates oxidative stress through the reduction of 105 lipid peroxidation products and that it has an immunomodulatory effect on cytokine secretion through increased cytokine secretion by the liver. cytokines through increased production of IFN-y and IL-l0, decreased production of IL-ly, stabilized tumor necrosis factor and secretion in HCV patients who have failed previous antiviral treatments.

Taking into account the benefits of Viusid, such as the reduction of inflammation and the immunomodulatory effect, a randomized double-blind study is proposed to evaluate the treatment with this food supplement in 200 patients with post-COVID syndrome diagnosed, assessing the improvement of their symptoms before and after treatment for 1 month, through clinical and paraclfnical examinations.

ELIGIBILITY:
Inclusion Criteria:

Patients with one or more of the following symptoms, persistent after suffering COVID-19:

* Extreme tiredness (Fatigue).
* Shortness of breath
* Chest pain
* Problems with memory or concentration ("Brain fog")
* Insomnia
* Palpitations
* Dizziness
* Tingling
* Joint pain
* Depression and anxiety
* Tinnitus or ear pain
* Malaise, diarrhea, stomach pain, loss of appetite
* Fever, cough, headache, dry throat, changes in sense of smell or taste
* Rash

Exclusion Criteria:

* Patients with a positive diagnosis of COVID-19 in the last 14 days.
* Patients who have presented symptoms similar to Post-COVID syndrome prior to the onset of COVID-19 due to a concomitant disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of the symptoms associated with post-COVID-19 syndrome. | 30 days
  Symptom assessment will be performed using the Visual Analogue Scale to Evaluate Fatigue Severity (VAS-F).
  The scale consists of 18 items relating to the subjective experience of fatigue. Each item asks respondents to place an "X," representing how they currently feel, along a visual analogue line that extends between two extremes. In contrast to discrete, Likert-type scales, the VAS-F places fewer restrictions on the range of responses available to individuals. However, the benefi ts of a visual analogue scale may be offset by the frequent reluctance of individuals to use the highest and lowest extremes.
  Scoring Each line is 100 mm in length - thus, scores fall between 0 and 100. The instrument also possesses two subscales: fatigue (items 1-5 and 11-18) and energy (items 6-10). Though individuals do not require training in order to score the scale, developers are quick to point out that high levels of inter-rater reliability are vital if results are to be correctly interpreted.
Evaluation of inflammation associated with Post-COVID-19 syndrome. | 30 days
  Evaluation of inflammation associated with Post-COVID-19 syndrome by analysis of IL-6 in venous blood samples before and after treatment, compared to the placebo group. The values for IL-6 concentration in the blood of healthy donors varied between 0 and 43.5 pg/ml. IL-6 concentrations above 43.5 pg/ml will be taken as inflammation values.
Evaluation of oxidative stress associated with Post-COVID-19 syndrome | 30 days
  Evaluation of oxidative stress associated with Post-COVID-19 syndrome by analysis of glutathione peroxidase concentration in venous blood samples before and after treatment, compared to the placebo group. Reference normal intervals range from 196 to 477 U/L in plasma, from 49 to 93 U/gHb in erythrocytes and from 52 to 96 U/gHb in whole blood.
Evaluation of pulmonar fibrosis associated with Post-COVID-19 syndrome | 30 days
  To evaluate the effect of Viusid on the recovery of respiratory symptoms associated with Post-COVID-19 syndrome by thoracic CT imaging analysis before and after treatment and in comparison with the placebo group.
  For the CT assessment, image analysis will be performed through digital processing, where different grayscale image data will be extracted in order to obtain numerical information about the evident pulmonary fibrosis, taking into account the intensity of the targets in the region of interest (i.e. lung tissue), comparing it with control images of healthy lungs. In addition, radiomic analysis and segmentation of the affected areas will be applied to obtain quantitative data on the severity of fibrosis. In addition, the images of interest will be visually analyzed by the project's medical staff, so that fibrosis can be directly diagnosed.

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación CR INVESTIGATION INSTITUTE, Bogotá, Bogotá DC, Colombia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] Montani D, Savale L, Noel N, Meyrignac O, Colle R, Gasnier M, Corruble E, Beurnier A, Jutant EM, Pham T, Lecoq AL, Papon JF, Figueiredo S, Harrois A, Humbert M, Monnet X; COMEBAC Study Group. Post-acute COVID-19 syndrome. Eur Respir Rev. 2022 Mar 9;31(163):210185. doi: 10.1183/16000617.0185-2021. Print 2022 Mar 31. PMID 35264409
- [Background] Silvagno F, Vernone A, Pescarmona GP. The Role of Glutathione in Protecting against the Severe Inflammatory Response Triggered by COVID-19. Antioxidants (Basel). 2020 Jul 16;9(7):624. doi: 10.3390/antiox9070624. PMID 32708578
- [Background] Sudre CH, Murray B, Varsavsky T, Graham MS, Penfold RS, Bowyer RC, Pujol JC, Klaser K, Antonelli M, Canas LS, Molteni E, Modat M, Jorge Cardoso M, May A, Ganesh S, Davies R, Nguyen LH, Drew DA, Astley CM, Joshi AD, Merino J, Tsereteli N, Fall T, Gomez MF, Duncan EL, Menni C, Williams FMK, Franks PW, Chan AT, Wolf J, Ourselin S, Spector T, Steves CJ. Attributes and predictors of long COVID. Nat Med. 2021 Apr;27(4):626-631. doi: 10.1038/s41591-021-01292-y. Epub 2021 Mar 10. PMID 33692530
- [Background] Vilar Gomez E, Gra Oramas B, Soler E, Llanio Navarro R, Ruenes Domech C. Viusid, a nutritional supplement, in combination with interferon alpha-2b and ribavirin in patients with chronic hepatitis C. Liver Int. 2007 Mar;27(2):247-59. doi: 10.1111/j.1478-3231.2006.01411.x. PMID 17311621